CLINICAL TRIAL: NCT01890213
Title: A Pilot Study of Active Immunotherapy With CEA(6D) VRP Vaccine (AVX701) in Patients With Stage III Colorectal Cancer
Brief Title: Immunotherapy With CEA(6D) VRP Vaccine (AVX701) in Patients With Stage III Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: AlphaVax, Inc. (Industry)
Responsible Party: Principal Investigator, Michael Morse, MD, Associate Professor, Duke University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00045976; IND13372 (Other: FDA)
Record Dates: First submitted 2013-06-26; First posted 2013-07-01 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Stage III Colon Cancer
Keywords: alphavirus; colon cancer; immune response; CEA
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vaccine (Experimental): AVX701 Vaccine:4 x 10EE8 IU intramuscularly every 3 weeks for 4 total immunizations
  Interventions: Biological: AVX701

INTERVENTIONS:
Biological: AVX701
  Other Names: VRP-CEA(6D)

SUMMARY:
This is a pilot study to evaluate the safety of a vaccine that consists of an alphavirus replicon (VRP) encoding the protein (CEA) that has been found to be associated with cancers such as colon cancer in patients that have stage III colon cancer. We will also evaluate the patient immune response to the vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage III colorectal cancer as determined by AJCC 7th edition.
* Subjects must have received adjuvant post-operative chemotherapy meeting the following requirements:

  1. Chemotherapy must have consisted of a 5-fluorouracil-based regimen with or without oxaliplatin for at least 6 cycles or capecitabine with or without oxaliplatin for 4 cycles.
  2. Chemotherapy must have been completed within 1-6 months of starting study treatment.
* Subjects with rectal cancer must have received chemotherapy meeting the following requirements:

  1. Neoadjuvant chemotherapy, if utilized, must have consisted of a 5-fluorouracil-based regimen (or capecitabine) with radiation
  2. Adjuvant chemotherapy must have consisted of a 5-fluorouracil-based regimen with or without oxaliplatin for at least 6 cycles or capecitabine with or without oxaliplatin for 4 cycles
  3. Chemotherapy must have been completed within 1-6 months of starting study treatment.
* Karnofsky performance status greater than or equal to 70%
* Estimated life expectancy > 6 months and not expected to require further systemic chemotherapy for at least 3 months.
* Age ≥ 18 years
* Adequate hematologic function: WBC ≥ 3000/microliter, Hgb ≥ 9 g/dL (may transfuse or use erythropoietin to achieve this level), platelets ≥ 100,000/microliter
* Adequate renal and hepatic function, with serum creatinine < 1.5 mg/dL, bilirubin < 1.5 mg/dL (except for Gilbert's syndrome which will allow bilirubin ≤ 2.0 mg/dL), ALT and AST ≤ 2.5 x upper limit of normal.
* Ability to understand and provide signed informed consent that fulfills Institutional Review Board's guidelines.
* Ability to return to Duke University Medical Center for adequate follow-up, as required by this protocol

Exclusion Criteria:

* Patients with active cytotoxic chemotherapy or radiation therapy should be excluded. There are no exclusions based on the number of prior chemotherapy, biologic, hormonal, or experimental regimens. There must be at least 3 months between any prior CEA-targeted immunotherapy and study treatment and at least 4 weeks between any other prior therapy and study treatment.
* Evidence of metastatic disease.
* Patients with a history of autoimmune disease, such as but not restricted to, inflammatory bowel disease, systemic lupus erythematosus, ankylosing spondylitis, scleroderma, or multiple sclerosis.
* Patients with serious intercurrent chronic or acute illness, such as cardiac disease (NYHA class III or IV), hepatic disease, or other illness considered by the Principal Investigator as unwarranted high risk for investigational drug treatment.
* Patients with a medical or psychological impediment to probable compliance with the protocol should be excluded.
* Concurrent (or within the last 5 years) second malignancy other than non melanoma skin cancer, cervical carcinoma in situ, or controlled superficial bladder cancer.
* Presence of an active acute or chronic infection including: a urinary tract infection , HIV (as determined by ELISA and confirmed by Western Blot) or viral hepatitis (as determined by HBsAg and Hepatitis C serology). Patients with HIV are excluded based on immuno-suppression, which may render them unable to respond to the vaccine; patients with chronic hepatitis are excluded because of concern that hepatitis could be exacerbated by the injections.
* Patients on steroid therapy (or other immuno-suppressives, such as azathioprine or cyclosporin A) are excluded on the basis of potential immune suppression. Patients must have had 6 weeks of discontinuation of any steroid therapy (except that used as pre-medication for chemotherapy or contrast-enhanced studies) prior to enrollment.
* Patients with allergies to any component of the vaccine will be excluded from the protocol.
* Pregnant and nursing women should be excluded from the protocol since this research may have unknown and harmful effects on an unborn child or on young children. If the patient is sexually active, the patient must agree to use a medically acceptable form of birth control while receiving treatment and for a period of 4 months following the last vaccination therapy. It is not known whether the treatment used in this study could affect the sperm and could potentially harm a child that may be fathered while on this study.
* Patients with acute or chronic skin disorders that will interfere with injection into the skin of the extremities or subsequent assessment of potential skin reactions will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2013-11 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Morse, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States